CLINICAL TRIAL: NCT00457964
Title: RAD001 Therapy of Angiomyolipomata in Patients With Tuberous Sclerosis Complex and Sporadic Lymphangioleiomyomatosis
Brief Title: RAD001 Therapy of Angiomyolipomata in Patients With TS Complex and Sporadic LAM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC IRB #2008-0812(04-07-22)
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Tuberous Sclerosis; Lymphangioleiomyomatosis
Keywords: Tuberous Sclerosis Complex (TSC); Lymyphangioleiomyomatosis; Mammalian Target of Rapamycin (mTOR); RAD001; Angiomyolipmas
MeSH Terms: conditions — Tuberous Sclerosis; Lymphangioleiomyomatosis; Hereditary Sensory and Autonomic Neuropathies | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Administration of RAD001 (Experimental)
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — 5 and 10 mg/day or 30, 50, 70mg/week

SUMMARY:
The purpose of this research study is to find out what effects RAD001 has on angiomyolipomas of a person with Tuberous Sclerosis Complex and to determine the safe dose of RAD001 without toxicity.

The hypothesis is that the drug will inhibit the growth of the angiomyolipomas and possibly even cause regression.

DETAILED DESCRIPTION:
Tuberous sclerosis complex is a genetic disorder with a birth incidence of approximately one in six thousand. Angiomyolipomas occur in eighty percent of persons with TS, and in up to 60% of persons with LAM. They are fatty tumors that often occur in kidney or liver as well as other parts of the body. They can grow and cause damage to surrounding kidney tissue and even renal failure. They may also leak blood causing potentially life-threatening hemorrhage.

Laboratory studies have shown that RAD001 suppresses the chemical that cause tumors to grow in tuberous sclerosis and sporadic LAM.

The primary goal of this study is to evaluate the clinical effectiveness of RAD001 in a 24 month trial. Although the primary goal is to determine if the drug RAD001 has effects on angiomyolipomas, other diseases associated with tuberous sclerosis will be monitored too, specifically any change in involvement of your brain or lungs with tuberous sclerosis. The use of RAD001 to treat angiomyolipomas in tuberous sclerosis or sporadic LAM is considered experimental

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with angiomyolipomas and have either Tuberous Sclerosis Complex or lymphangioleiomyomatosis
* Angiomyolipoma one centimeter or greater in largest diameter
* Between the ages of 18 and 65 years old.
* If female, documentation of negative pregnancy test prior to enrollment and, where applicable, use of appropriate non-estrogen containing birth control contraceptive regimen while on study.
* Adequate renal function (creatinine < 3 mg/dl)

Exclusion Criteria:

* Pregnant or lactating women
* Continuous requirement for supplemental oxygen
* Surgery within past 2 months
* Use of an investigational drug within last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Patients will be considered responders if their angiomyolipoma volume decreases by thirty percent or more from baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John J. Bissler, M.D., Principal Investigator — LaBonheur Children's Hospital
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States